CLINICAL TRIAL: NCT00452881
Title: A Randomized Phase II Study Adjuvant Gemcitabine And Oxaliplatin Versus Gemcitabine and Cisplatin for Completely Resected Stage IB, II or IIIA Non-Small Cell Lung Cancer
Brief Title: Adjuvant Gemcitabine Plus Oxaliplatin Versus Gemcitabine Plus Cisplatin for Completely Resected Stage IB/II/IIIA NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-158
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
Keywords: Non-small cell lung cancer; adjuvant chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Oxaliplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study arm (Experimental): GemOx
  Interventions: Drug: gemcitabine; Drug: Oxaliplatin
- control arm (Active Comparator): GemCis
  Interventions: Drug: gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: gemcitabine — Gemcitabine1250mg/m2 iv on day 1 and 15, every 4weeks, maximum 4 cycles
Drug: Oxaliplatin — Oxaliplatin 85mg/m2 iv on day 1 and 15, every 4 weeks, maximum 4 cycles
  Arms: study arm
Drug: Cisplatin — Cisplatin 40mg/m2 iv on day 1 and 15, every 4 weeks, maximum 4 cycles
  Arms: control arm

SUMMARY:
Oxaliplatin has a more manageable toxicity profile than cisplatin, with no renal toxicity and a lower incidence of hematological and gastrointestinal toxicities. The combination of gemcitabine-oxaliplatin is attractive in NSCLC patients as it may improve the therapeutic index. Given the potential advantages of oxaliplatin and th finding that the addition of chemotherapy improves survival in the postoperative adjuvant setting, we conduct a phase II trial to compare adjuvant gemcitabine-oxaliplatin with gemcitabine-cisplatin in patients with completely resected stage IB, II or IIIA NSCLC

DETAILED DESCRIPTION:
This study is a randomized phase II study. Patients are randomized to 1 of 2 treatment arms: patients receive adjuvant chemotherapy with gemcitabine-oxaliplatin or gemcitabine-cisplatin. Chemotherapy should be started within 8 weeks after complete surgical resection. Patients are followed every 3 months for 2 years, every 6 months for 3 years.

Gemcitabine-Oxaliplatin (GemOx) chemotherapy:

Gemcitabine (1,250 mg/m2)+Oxaliplatin (85 mg/m2) is given on day 1 and 15 q 4weeks. maximum 4 cycles.

Gemcitabine-Cisplatin (GemCis) chemotherapy:

Gemcitabine (1,250 mg/m2) + Cisplatin (40 mg/m2) is given on day 1 and 15 q 4weeks. maximum 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of non-small cell lung cancer.
2. Presence of pathological stage IB, II or IIIA, according to the American Joint Committee on Cancer (AJCC).
3. Completely resected tumor at NCC hospital.
4. No prior tumor therapy (radiotherapy, chemotherapy, immunotherapy, or any other type of tumor therapy).
5. Performance status of 0-1 on ECOG scale.
6. At least 18 years old
7. Patient compliance that allows adequate follow-up.
8. Adequate organ function including the following:Adequate hematologic function: WBC count ≥ 4,000/uL, absolute neutrophil count (ANC) ≥ 1,500/uL, platelet count ≥ 100,000/uL, and hemoglobin ³ 10 gm/dL.Adequate hepatic function: bilirubin ≤ 1.5 x UNL, ALT or AST ≤ 2.5 x UNL.Adequate renal function: creatinine ≤ 1.5mg/dL.
9. Signed informed consent from patient or legal representative.
10. Patients with reproductive potential must use an approved contraceptive method during and for 3 months after the study. Females with childbearing potential must have a negative urine hCG test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Concurrent administration of any other tumor therapy, including radiotherapy, chemotherapy, immunotherapy.
2. Active uncontrolled infection.
3. Serious concomitant disorders that would compromise the safety of patient or compromise the patient's ability to tolerate therapy.
4. Second primary malignancy.
5. Significant neurological or mental disorder.
6. Pregnant or nursing.
7. MI within preceding 6 months or symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Compare time to recurrence with these regimens | the first day of the treatment to date of the tumor recurrence

SECONDARY OUTCOMES:
Compare to Overall survival with these regimens | the first day of treatment to death
Compare to Toxicities with these regimens | the first day of treatment to the date that disease progression is reported
- To define the patient population most at risk for disease recurrence | from the date of randomization to date of recurrence
(tissue banking and blood sampling for analysis of predictive markers) | before treatment, obtained from the resected lung cancer specimen
Compare quality of life as assessed by EORTC QLQ-C30, EORTC QLQ-LC13 with these regimens | before treatment and after each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Ill Zo, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea